CLINICAL TRIAL: NCT04853693
Title: Pregnancy Without Psychosocial Stress - the Earliest Prevention of Mental Disorders and Toxic Stress in Children
Brief Title: Pregnancy Without Psychosocial Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZD-ZDOVA1-018
Record Dates: First submitted 2021-04-08; First posted 2021-04-21 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Depressive Symptoms; Anxiety Disorders and Symptoms; Depression, Postpartum
MeSH Terms: conditions — Depression; Anxiety Disorders; Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Two groups: One receives MSM prevention intervention and the other group receives Enhanced Treatment as Usual (referral and monitoring).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and person administering the outcome measures are blind to participant group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mom´s Supporting Mom (MSM) (Experimental): A preventive intervention that involves psychoeducation and peer techniques described in study detailed description.
  Interventions: Behavioral: Mom´s Supporting Mom
- Enhanced Treatment as Usual (Active Comparator): Referral to treatment in the community and monitoring
  Interventions: Behavioral: Enhanced Treatment As Usual

INTERVENTIONS:
Behavioral: Mom´s Supporting Mom — A preventive peer consultation intervention for Postpartum Depression.
  Other Names: MSM
  Arms: Mom´s Supporting Mom (MSM)
Behavioral: Enhanced Treatment As Usual — Referral to treatment in the community, clinical monitoring
  Other Names: ETAU
  Arms: Enhanced Treatment as Usual

SUMMARY:
The project is aimed at children who are exposed to the toxic psychosocial stress present in their mothers during pregnancy or after childbirth. Due to psychosocial stress in their mothers, these children are at risk of developing a mental disorder or having impaired psychosocial development.

In Czechia, there is no prevention of psychosocial stress in women, which also plays a preventive role in the development of mental disorders in their children. Mental disorders in parents are stigmatized in Czechia, which prevents parents from seeking care.

The investigators want to change this situation, so they will:

1. create and pilot a screening program for psychosocial stress in perinatal women in gynecological clinics
2. connect the screening program to the integrated step care system created by the investigators, including peer support, which the investigators will test

DETAILED DESCRIPTION:
ACTIVITY 1 Objective of the activity: To increase the support of mental health and well-being of unborn children and children in the period soon after their birth by early detection of women experiencing psychosocial stress during pregnancy and after childbirth. Target group: Pregnant women and postpartum women and their children.

Methods: Because the occurrence of symptoms of psychosocial stress in pregnancy is one of the main predictors of the development of mental disorders after childbirth, the investigators will test whether the introduction of screening in gynecological clinics during pregnancy reduces the incidence of untreated mental disorders in women 6 weeks after birth. Thanks to screening, the investigators want to capture women and their children who are exposed to toxic stress during pregnancy. Screening: Gynecological clinics will be equipped with a tablet with screening software (Czech version of the Edinburgh Perinatal Depression Scale; Perinatal Anxiety Screening Scale; Perinatal Psychosocial Profile). The software runs on the servers of the National Institute of Mental Health (NUDZ), secured against cybercrime. Work with data obtained during screening is subject to GDPR and the process is approved by the NUDZ Ethics Committee. The screening software is automated and sends the woman information about the results to her email.

Evaluation: a randomized controlled study in 20 gynecological clinics in 3 regions of the Czech Republic (Prague, Central Bohemia and Olomouc Region). Participating gynecological outpatient clinics will be randomized in a 1: 1 ratio into two groups: Intervention outpatient clinics: Intervention outpatient clinics offer study participation to all pregnant women during their pregnancy. Furthermore, all women checked at the end of the sixth week. Intervention clinics will also be equipped with information materials on mental health during pregnancy and after childbirth. Control clinics: actively offer participation to all women only at the control at the end of the sixth week postpartum. The main checkpoint in both groups of outpatient clinics is the 6th week after delivery, when the woman comes to the gynecological outpatient clinic for a mandatory check-up in Czechia. All women who will participate in Activity 1 will be examined by telephone using a structured psychiatric examination by a psychiatrist at the end of the 6th week after childbirth so that we can determine the presence of mental disorders.

Hypothesis: There are more women in control clinics who are not treated for a mental disorder at the end of the 6th week after delivery, even if they have been diagnosed, than in intervention clinics.

ACTIVITY 2 Objective of the activity: To increase the support of mental health and well-being of unborn children and children soon after their birth through early intervention in women experiencing psychosocial stress during pregnancy and after childbirth. Target group: Women who experience psychosocial stress during pregnancy and after childbirth and their children. Methods: Activity 2 is directly related to activity 1 of the submitted project. As part of Activity 2, the investigators will provide the women captured by the screening intervention developed by them.

Intervention: Mom supports Mom includes at least four telephone or other contacts - Skype, Zoom, WhatsApp, Facebook Messenger, ...) Between the project participant and a peer consultant trained by the National Institute of Mental Health and Mom´s Smile. Within peer support, the main methods are listening, psychoeducation, basic procedures of cognitive behavioral therapy and mindfulness, shared personal experiences with perinatal psychosocial stress and, if necessary, a reference to professional counseling (psychology, psychiatry).

Evaluation: a randomized controlled study in gynecological clinics participating in Activity 1 of the project. Women experiencing psychosocial stress, which we will screen through Activity 1, will be randomized 1: 1 into two groups: Intervention group: The peer consultant coordinator will connect the woman with the peer consultant who will carry out the intervention Mom supports mom. Control group: The woman will be sent automatic feedback with information on how to proceed if the participant wants to seek help herself. Evaluation of the effect of the intervention: The investigators evaluate depressive symptoms using the Edinburgh scale of perinatal depression; anxiety symptoms using the Perinatal Anxiety Screening Scale; psychosocial stress using the Perinatal Psychosocial Profile; quality of life using the 8-dimensional quality of life scale; and parental competences using the Parenting Sense of Competence Scale. The investigators collect data after the woman enters Activity 2 and one month after entering. The Investigators will evaluate the feedback from users using qualitative questions.

Hypothesis: Intervention Mom supports mom, reduces depressive and anxiety symptoms and general psychosocial stress in women experiencing psychosocial stress. Intervention Mom supports mom, increases the quality of life and parental competencies of women experiencing psychosocial stress.

Statistics: n = 120 (60 in each arm of the study). Sample size is calculated so that the investigators can detect a medium-to-large group difference in the scale of depressive symptoms (effect size = 0.6; t-test) at power 80%, significance level 5% (2-sided) and potential drop out 30 %.

ELIGIBILITY:
Inclusion Criteria ACTIVITY 1:

* sex-female
* pregnancy
* woman is registered during and after pregnancy in one of 20 study gynecological outpatient clinics
* signing informed consent
* email address ownership
* age 18-45

Inclusion Criteria ACTIVITY 2:

* Edinburgh Postpartum Depression Scale score ≥10.
* participant identified through the ACTIVITY 1 of the study

Exclusion Criteria ACTIVITY 1:

- acute medical illness or significant pregnancy complication (based on self-report)

Exclusion Criteria ACTIVITY 2:

* acute suicidal behavior (based on self-report)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment gap for postpartum mental disorders | 6 weeks postpartum
  prevalence of untreated mental health disorders in postpartum women assessed by The Mini-International Neuropsychiatric Interview
Pregnancy depressive symptoms | up to 32 weeks
  self-rated depressive symptomatology measured by Edinburgh Postnatal Depression Scale. Score range 0-30, higher score represents worse outcome.
Postpartum depressive symptoms | 6 weeks postpartum
  self-rated depressive symptomatology measured by Edinburgh Postnatal Depression Scale. Score range 0-30, higher score represents worse outcome.

SECONDARY OUTCOMES:
Pregnancy anxiety symptoms | up to 32 weeks
  self-rated anxiety symptomatology measured by Perinatal Anxiety Screening Scale. Score range 0-93, higher score represents worse outcome.
Postpartum anxiety symptoms | 6 weeks postpartum
  self-rated anxiety symptomatology measured by Perinatal Anxiety Screening Scale. Score range 0-93, higher score represents worse outcome.

OTHER OUTCOMES:
Psychosocial stress factors | through study completion, an average of 1 year
  self-rated psychosocial stress factors measured by Prenatal psychosocial profile. Score range 11 - 44, higher score represents worse outcome.
Prenatal mother-baby attachment | up to 32 weeks
  self-report measure of maternal-fetal attachment measured by Prenatal Attachment Inventory
Parenting competences | 6 weeks postpartum
  self-report measure od maternal sense of parenting competence measured by Parenting Sense of Competence Scale

CONTACTS AND LOCATIONS:
Overall Officials: Antonin Sebela, Ph.D., Principal Investigator — National Institute of Mental Health, Klecany, Czechia
Locations (1):
- National Institute of Mental Health, Klecany, Czechia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be made available to other researchers.
Supporting Information: ICF
Time Frame: After the completion of the study
Access Criteria: Permission of the PI

REFERENCES:
- [Derived] Horakova A, Kuklova M, Hrdlickova K, Nemcova H, Knytl P, Kostylkova L, Sebela A. Effectiveness of the mom supports mom peer support intervention in treating antenatal mental health difficulties in women. Midwifery. 2024 Dec;139:104198. doi: 10.1016/j.midw.2024.104198. Epub 2024 Sep 24. PMID 39342905